CLINICAL TRIAL: NCT04520386
Title: A Multi-site, Single Arm, Phase II Clinical Trial, to Evaluate the Efficacy of OMT-111 in Supporting the Treatment of Terminal Stage Solid Tumors
Brief Title: OMT-111 for Terminal Stage Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MetiMedi Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Metimedi-202
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Pancreatic Cancer; Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label single arm (Experimental): 1 cycle consists of 4 weeks (28 days). Each week consists of 5 days of treatment and 2 days of treatment-free interval
  Interventions: Drug: OMT-111

INTERVENTIONS:
Drug: OMT-111 — Pre-filled Syringe
  Other Names: OMT-110

SUMMARY:
Patients with terminal stage of metastatic non-small cell lung cancer, metastatic triple negative breast cancer, or advanced or metastatic pancreatic adenocarcinoma resisting to standard therapies.

DETAILED DESCRIPTION:
This is a multi-site, single arm, Phase II study designed to explore the efficacy of OMT-111 in patients with terminal stage solid tumors resistant to standard therapies.

Subjects who voluntarily provide written consent to participate in this study undergo screening tests within 4 weeks prior to the first dose of investigational product. Those who meet the inclusion/exclusion criteria are enrolled in the study.

1 cycle consists of 4 weeks (28 days). Each week consists of 5 days of treatment and 2 days of treatment-free interval (20 days of treatment and 8 days of treatment-free interval per cycle in total). This study is planned to enroll approximately 76 subjects including 42 subjects with lung cancer, 22 subjects with breast cancer, and 12 subjects with pancreatic cancer. Treatment will be provided for 12 cycles (48 weeks). During the study, tests and procedures to evaluate the efficacy and safety will be carried out according to the planned schedule.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer

  1. Female at least 18 years old or older at the time of informed consent
  2. Histologically or cytologically confirmed triple negative ductal adenocarcinoma of breast
  3. Patients who have visceral metastatic lesions not amenable by resection or radiotherapy (e.g., multiple visceral lesions)
  4. ECOG PS (Eastern Cooperative Oncology Group Performance Status): 0-2
  5. Patients with a life expectancy ≥ 12 weeks as judged by the investigator
  6. At least one measurable lesion or evaluable lesion defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Pancreatic Cancer

  1. Male or female at least 18 years old or older at the time of informed consent
  2. Histologically or cytologically confirmed adenocarcinoma of pancreas
  3. Patients who have advanced or metastatic lesions not amenable by resection or radiotherapy
  4. ECOG PS (Eastern Cooperative Oncology Group Performance Status) ≤ 2
  5. Patients with a life expectancy ≥ 12 weeks as judged by the investigator
  6. At least one measurable lesion or evaluable lesion defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Lung Cancer

  1. Male or female at least 18 years old or older at the time of informed consent
  2. Histologically or cytologically confirmed carcinoma of the lung (small cell lung cancer not included)
  3. Patients who have unresectable metastatic lesion
  4. ECOG PS (Eastern Cooperative Oncology Group Performance status) ≤ 2
  5. Patients with a life expectancy ≥ 12 weeks as judged by the investigator
  6. At least one measurable lesion or evaluable lesion defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

Exclusion Criteria:

* Breast Cancer

  1. History of malignancy other than metastatic triple negative breast cancer within 5 years prior to the first dose of investigational product (however, patients with effectively treated skin cancer, thyroid cancer, and carcinoma in situ that has been in complete remission for at least 3 years and thus considered cured by the investigator are eligible)
  2. Uncontrolled CNS metastasis (however, patients with treated and stable brain metastasis (radiographically stable for at least 30 days without steroids) are eligible)
  3. Primary cancer-related complications potentially requiring urgent surgery as judged by the investigator
  4. Grade ≥ 3 active infection requiring intravenous antibiotics per NCI-CTCAE version 5.0
  5. History of one or more of the following cardiovascular diseases

     * Cerebrovascular disease, unstable angina, or myocardial infarction within 6 months prior to the screening visit (Visit 1)
     * Congestive heart failure corresponding to New York Heart Association (NYHA) Class III or above (see Appendix 1. NYHA Classification)
     * Serious cardiac arrhythmia not controlled with medication or clinically significant cardiovascular abnormality as judged by the investigator
     * QTc > 480 msec (Fredericia's formula) during 12-lead ECG at screening visit (Visit 1)
  6. Pregnant women, breast-feeding women or women with a positive pregnancy test at screening visit (Visit 1)
  7. Renal impairment or chronic renal failure patient requiring hemo- or peritoneal dialysis
  8. Previous treatment with the investigational product
  9. Treatment with other investigational product within 30 days prior to the first dose of the investigational product
  10. Unable to come to the site hospital on a daily basis for investigational product administration
  11. Patients who are otherwise considered to be ineligible for this study based on investigator's judgment.
* Pancreatic Cancer

  1. History of malignancy other than advanced or metastatic pancreatic adenocarcinoma within 5 years prior to the first dose of investigational product (however, patients with effectively treated skin cancer, thyroid cancer, and carcinoma in situ that has been in complete remission for at least 3 years and thus considered cured by the investigator are eligible)
  2. Uncontrolled CNS metastasis (however, patients with treated and stable brain metastasis (radiographically stable for at least 30 days without steroids) are eligible)
  3. Primary cancer-related complication potentially requiring urgent surgery as judged by the investigator
  4. Grade ≥ 3 active infection requiring intravenous antibiotics per NCI-CTCAE version 5.0
  5. History of one or more of the following cardiovascular diseases

     * Cerebrovascular disease, unstable angina, or myocardial infarction within 6 months prior to the screening visit (Visit 1)
     * Congestive heart failure corresponding to New York Heart Association (NYHA) Class III or above (see Appendix 1. NYHA Classification)
     * Serious cardiac arrhythmia not controlled with medication or clinically significant cardiovascular abnormality as judged by the investigator
     * QTc > 480 msec (Fredericia's formula) during 12-lead ECG at screening visit (Visit 1)
  6. Pregnant women, breast-feeding women or women with a positive pregnancy test at screening visit (Visit 1)
  7. Renal impairment or chronic renal failure patient requiring hemo- or peritoneal dialysis
  8. Previous treatment with the investigational product
  9. Treatment with other investigational product within 30 days prior to the first dose of the investigational product
  10. Unable to come to the site hospital on a daily basis for investigational product administration
  11. Patients who are otherwise considered to be ineligible for this study based on investigator's judgment
* Lung Cancer

  1. History of malignancy other than metastatic non-small cell lung cancer within 5 years prior to the first dose of investigational product (however, patients with effectively treated skin cancer, thyroid cancer, and carcinoma in situ that has been in complete remission for at least 3 years and thus considered cured by the investigator are eligible)
  2. Uncontrolled CNS metastasis (however, patients with treated and stable brain metastasis (radiographically stable for at least 30 days) are eligible)
  3. Primary cancer-related complication potentially requiring urgent surgery as judged by the investigator
  4. Grade ≥ 3 active infection requiring intravenous antibiotics per NCI-CTCAE version 5.0
  5. History of one or more of the following cardiovascular diseases

     * Cerebrovascular disease, unstable angina, or myocardial infarction within 6 months prior to the screening visit (Visit 1)
     * Congestive heart failure corresponding to New York Heart Association (NYHA) Class III or above (see Appendix 1. NYHA Classification)
     * Serious cardiac arrhythmia not controlled with medication or clinically significant cardiovascular abnormality as judged by the investigator
     * QTc > 480 msec (Fredericia's formula) during 12-lead ECG at screening visit (Visit 1)
  6. Pregnant women, breast-feeding women or women with a positive pregnancy test at screening visit (Visit 1)
  7. Renal impairment or chronic renal failure patient requiring hemo- or peritoneal dialysis
  8. Previous treatment with the investigational product
  9. Treatment with other investigational product within 30 days prior to the first dose of the investigational product
  10. Unable to come to the site hospital on a daily basis for investigational product administration
  11. Patients who are otherwise considered to be ineligible for this study based on investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | From the start of treatment to 48 weeks.
  Every two cycles (8 weeks)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the start of treatment to 48 weeks.
  Every two cycles (8 weeks)
Duration of Response (DoR) | From the start of treatment to 48 weeks.
  Every two cycles (8 weeks)
Progression-Free Survival (PFS) | From the start of treatment to 48 weeks.
  Every two cycles (8 weeks)
18F-FDG- PET/CT (SUVmean and SUVmax) | From the start of treatment to 48 weeks.
  Every two cycles (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Soobong Park, Study Director — MetiMedi Pharmaceuticals
Locations (2):
- Vietnam (2):
  - K Hospital, Hanoi
  - Cho Ray Hospital, Hochiminh City

IPD SHARING:
Plan to Share IPD: No